CLINICAL TRIAL: NCT04727515
Title: General Anesthesia, Versus Axillary Block for Ambulatory Hand Surgery: Randomized Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mennatullah Mohammed, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU M D 186/2019
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Fentanyl; Isoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Experimental): Patients will receive general anesthesia
  Interventions: Drug: fentanyl 2µg/kg intravenously and maintained with isoflurane
- Axillary Block (Experimental): Patients will receive axillary nerve block
  Interventions: Procedure: Axillary nerve Block

INTERVENTIONS:
Drug: fentanyl 2µg/kg intravenously and maintained with isoflurane — Anesthesia will be induced using titration of intravenous propofol till loss of verbal contact and fentanyl 2µg/kg intravenously and maintained with isoflurane (end tidal up to 1.5%), oxygen in air 50:50 via a laryngeal mask.
  Arms: General anesthesia
Procedure: Axillary nerve Block — Axillary block will be performed using ultrasound technique. Patients will receive an axillary block under ultrasound guidance using a linear 5-12 MHz probe.
  Arms: Axillary Block

SUMMARY:
This study aims to compare between general anesthesia and axillary nerve block for ambulatory hand surgery regarding postoperative sleep pattern and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Physical Status: ASA I and II Patients after taking written and informed consent
* Body mass index less than 30

Exclusion Criteria:

* Refusal of procedure or participation in the study by patients.
* Physical status: ASA III or above
* Subjects presenting with allergy to local anesthetics, alcohol or drug abuse.
* Inability to cooperate mentally retarded patients.
* Bleeding disorders.
* Patients with preoperative obstructive sleep apnea (OSA) or any sleep disturbance.
* Patients with body mass index more than 30.
* Polytrauma patients or emergency operation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative nausea and vomiting | First 24 hours postoperatively
  Incidence of postoperative nausea and vomiting requiring treatment

SECONDARY OUTCOMES:
Visual analogue scale [VAS] | First 24 hours postoperatively
  Visual analogue scale [VAS] will be used to measure pain score at 30 min, 1, 2, 4, 6, 8, 10, 12 and 24 h after surgery. All the study patients will be instructed about the use of the VAS scale before induction of anesthesia (VAS score 0 cm = no pain, VAS score 10 cm = worst possible pain)
Pittsburgh Sleep Quality Index | First 24 hours postoperatively
  Pittsburgh Sleep Quality Index will be used to measure postoperative sleep disturbance. It is formed of 19 items that assess seven clinically derived domains of sleep difficulties (Sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction) over a Likert scale (0-3)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt